CLINICAL TRIAL: NCT06053658
Title: Phase 2 Study of Combination Tivozanib and Nivolumab in Advanced Non-Clear Cell Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0485; NCI-2023-07385 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — tivozanib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Tivozanib and Nivolumab (Experimental): Nivolumab by vein over about 60 minutes every 4 weeks (Day 1 of each cycle). Tivozanib tablets by mouth 1 time every day for 21 days (Days 1-21 of each cycle), and then no tablets on Days 22-28 of each cycle.
  Interventions: Drug: Tivozanib; Drug: Nivolumab

INTERVENTIONS:
Drug: Tivozanib — Given by PO
  Other Names: KRN 951; KRN-951; KRN951; UNII-172030934T; AV951; AV951 cpd
Drug: Nivolumab — Given by IV (vein)
  Other Names: Opdivo; BMS-936558

SUMMARY:
To learn if giving tivozanib in combination with nivolumab can help to control advanced nccRCC.

DETAILED DESCRIPTION:
Primary Objectives

* To demonstrate efficacy of combination tivozanib and nivolumab in advanced non-clear cell renal cell carcinoma (nccRCC).

Secondary Objectives

* To assess the safety and toxicity of combination tivozanib and nivolumab.
* To estimate the duration of clinical efficacy

Exploratory Objectives

* To associate immune and tumor biomarkers with clinical efficacy

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed metastatic non-clear cell renal cell carcinoma of papillary, chromophobe, oncocytic neoplasms, unclassified, or not otherwise specified (NOS) as clear cell. Medullary carcinoma of the kidney and collecting duct tumors are NOT allowed
2. Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
3. Up to 1 systemic line of therapy (either monotherapy or combination) including prior immunotherapy (anti-PD1, PD-L1, or CTLA-4) and multi-tyrosine kinase inhibitors in non-metastatic or metastatic setting is allowed. A washout period of 5 half lives or 21 days, whichever one is shorter, will be required for patients that have received previous systemic therapy.
4. Age ≥18 years.
5. Eastern Cooperative Oncology Group (ECOG) Appendix 1 performance status ≤2 (Karnofsky ≥60%).
6. Patients must have adequate organ and marrow function as defined below:

   1. absolute neutrophil count ≥1,000/mcL
   2. platelets ≥100,000/mcL
   3. total bilirubin ≤ institutional upper limit of normal (ULN)
   4. AST ≤3 × institutional ULN
   5. (ALT) ≤3 × institutional ULN
   6. creatinine ≤1.5 × institutional ULN
   7. eGFR ≥30 ml/min
7. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
8. For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
9. Patients with treated brain metastases (at least 4 weeks have passed from treatment) are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.
10. Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy.
11. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
12. Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
13. The effects of combination tivozanib and nivolumab on the developing human fetus are unknown. For this reason and because tyrosine kinase inhibitors and immunotherapy agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (refer to MDA Policy CLN 1114) This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

    * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
    * History of hysterectomy or bilateral salpingo-oophorectomy.
    * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
    * History of bilateral tubal ligation or another surgical sterilization procedure. Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device, Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide.

    Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
14. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of combination tivozanib and nivolumab administration.
15. Participants or their legally acceptable representative (LAR) must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal participant care.

Exclusion Criteria:

1. Prior tivozanib therapy.
2. Prior nivolumab therapy.
3. Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
4. Patients who are receiving any other investigational agents.
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition to tivozanib or nivolumab.
6. Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg on 2 or more antihypertensive medications, documented on 2 consecutive measurements taken at least 2 hours apart. Anti-hypertensives must not have been increased 30 days prior to enrollment.
7. History of autoimmune disorders except for the following:

   1. Patients with vitiligo or alopecia
   2. Hypothyroidism (e.g. following Hashimoto syndrome) that is stable on thyroid hormone replacement
   3. Any chronic skin condition that does not require systemic therapy
   4. Patients without active autoimmune disease requiring treatment in the last 3 years may be included after consultation with study MDA lead Principal Investigator
8. Active human immunodeficiency virus (HIV) infection unless patients are on effective anti-retroviral therapy with undetectable viral load within 6 months.
9. Has evidence of any other medical conditions, psychiatric condition, physical examination or laboratory findings that may interfere with the planned treatment, affect subject compliance or place the subject at high risk from treatment-related complications in the opinion of the local principal investigator (PI).
10. Current systemic corticosteroid use greater than prednisone 10 mg daily or equivalent.
11. Pregnant women are excluded from this study because tivozanib and nivolumab are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with tivozanib and nivolumab, breastfeeding should be discontinued if the mother is treated with tivozanib and nivolumab.
12. Receiving concomitant CYP3A inducers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jonasch, M D, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - UT Southwestern Medical Center, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT06053658/ICF_000.pdf